CLINICAL TRIAL: NCT06096805
Title: Prediction of Placental Fetal Growth Restriction in High Risk Population (PoPFGR)
Status: Recruiting | Type: Observational
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Luming Sun, Professor, Shanghai First Maternity and Infant Hospital
Other Study IDs: ShanghaiFMIH-FMU7
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — maternal blood, urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to prospectively enroll high-risk pregnant women to establish a multicenter cohort. By combining maternal basic characteristics, medical history, early pregnancy ultrasound, and biological markers, we aim to construct a joint predictive model for MVM-FGR.

DETAILED DESCRIPTION:
Clinical guidelines do not recommend clinical screening for MVM-FGR in low-risk populations. Predictive models for FGR are often based on preeclampsia prediction models or Down syndrome serum screening models, which have limited utility. This study aims to establish a multi-center prospective cohort of pregnant women at high risk for FGR. We will collect baseline characteristics of pregnant women, ultrasound measurements of fetal growth, structural scans, maternal-fetal Doppler blood flow, as well as maternal serum and plasma in first and mid-trimester. Serum and plasma biomarker testing will be conducted. We will regularly observe fetal growth data, maternal-fetal complications during pregnancy, and collect delivery information, conditions of the newborn and placental pathology results after birth. By integrating maternal medical history, serum and plasma biomarkers, Doppler ultrasound, and other factors, we will establish a combined predictive model for early and mid-term MVM-FGR.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestational age of <14 weeks
* Maternal age between 18 and 45 years old
* With at least one of FGR high risk factors:

  1. Maternal age >40 years
  2. Nulliparous, Maternal age >38 years
  3. Previous pregnancy with FGR, PE or placental abruption
  4. Maternal medical history of chronic hypertension, diabetes mellitus, chronic nephritis or autoimmune diseases (such as SLE or APS)
  5. Recurrent spontaneous abortion (RSA) > 3 times with unknown causes
* Or with at least two of the following FGR high risk factors:

  1. Maternal age 35~40 years
  2. BMI ≥ 28 kg/m2 or BMI < 18.5 kg/m2
  3. Conception with assisted reproductive technology
  4. Interval from previous delivery: > 5 years or < 6 months

     Exclusion Criteria:
* Presence of fetal genetic abnormalities or severe structural abnormalities in prenatal ultrasound or genetic testing.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — First trimester pregnancy women who are at higher risk of fetal growth restriction.
Study Population: First trimester pregnancy women who are at higher risk of fetal growth restriction.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Present of maternal-vascular-malperfusion (MVM)-FGR | during the pregnancy, up to an average gestational age of 40 weeks
  Development of MVM Fetal growth restriction

SECONDARY OUTCOMES:
Other adverse pregnancy outcome | pregnancy-born after 28 days
  including miscarriage, preeclampsia; intrauterine fetal death
GA at delivery, birth weight, neonatal outcomes. | the day at birth
  GA at delivery, birth weight, neonatal outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Luming Sun, Docter, Principal Investigator — Shanghai First Maternity and Infant Hospital
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China